CLINICAL TRIAL: NCT01344785
Title: The Effect of Loss of Offset After Pertrochanteric Fracture Treated With a Intramedullary Nail
Acronym: PLAIN
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Consultant Orthopaedic surgeon, Danderyd Hospital
Other Study IDs: PLAIN-1
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Intertrochanteric Fractures
Keywords: Intertrochanteric Fractures; Intramedullary nailing; Hip function; Pain
MeSH Terms: conditions — Hip Fractures; Pain | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a intertrochanteric fracture: Patients with a intertrochanteric fracture, n=100
  Interventions: Procedure: Intramedullary nailing

INTERVENTIONS:
Procedure: Intramedullary nailing — All patients will be treated with Intramedullary nailing
  Other Names: Gamma 3, Stryker, USA

SUMMARY:
The purpose of this study is determine the relationship between pain and protrusion of the implant after surgery for a intertrochanteric fracture.

DETAILED DESCRIPTION:
Intertrochanteric fractures are common fractures in which severe complications such as non-union, implant cut-out and postoperative wound-infections occur at very low rates with modern surgical techniques. While severe complications are rare, the patient reported outcome is less satisfactory with roughly half of the patients complain of thigh pain and others failing to regain their walking ability. The current leading methods for osteosynthesis of intertrochanteric fractures are intramedullary (IM) nails and sliding hip screws (SHS).

Over the period 1998 to 2007 the use of IM nails for pertrochanteric fractures increased from 5% to 20% in Sweden, at the expense of the use of SHS (5). IM nailing has also become more common at our clinic where we since February 2008 use the 3rd generation of the Gamma nail. In this study we investigate if the increased pain after IM nailing, reduced hip function and life quality may correlate to the compression over the fracture and the lateral protrusion of the intramedullary nail.

ELIGIBILITY:
Inclusion Criteria:

* Intertrochanteric Fracture
* Age over 55
* Intramedullary nailing

Exclusion Criteria:

* Severe cognitive impairment
* Substance abuse

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 consecutive patients with an intertrochanteric fracture presenting at the Orthopaedic depertment of Danderyd Hospital, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Hip function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Max Gordon, MD, Principal Investigator — Danderyd Hospital
Locations (1):
- Danderyd Hospital, Stockholm, Sweden